CLINICAL TRIAL: NCT01431352
Title: The Effects of Chinese Herbal Medicine and Letrozole on Live Birth in Infertile Women With Polycystic Ovary Syndrome:A Double-blind Randomized Controlled Trial
Brief Title: Letrozole Versus Chinese Herbal Medicine on Polycystic Ovary Syndrome (PCOS)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Heilongjiang University of Chinese Medicine (Other)
Responsible Party: Principal Investigator, Xiaoke Wu, Professor and Chairman Dept Obs & Gyn, First Affiliated Hospital, Heilongjiang University of Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Letrozole
Record Dates: First submitted 2011-09-06; First posted 2011-09-09 (Estimated); Last update posted 2013-11-05 (Estimated); Status verified 2013-11

CONDITIONS: Polycystic Ovary Syndrome
Keywords: Polycystic ovary syndrome; Randomized controlled trial; Chinese herbal medicine; Chinese herbal medicine granules; Letrozole; Live birth
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Letrozole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Letrozole+ Chinese herbal medicine granules (Experimental)
  Interventions: Drug: Letrozole; Drug: Chinese herbal medicine granules or Chinese herbal medicine granules placebo
- Letrozole+ Chinese herbal medicine granules placebo (Placebo Comparator)
  Interventions: Drug: Letrozole

INTERVENTIONS:
Drug: Letrozole — 2.5 mg letrozole daily from day 5 of the menses for 5 days for month 1 to 3, 5.0 mg letrozole daily from day 5 of the menses for 5 days for month 4 to 6.
Drug: Chinese herbal medicine granules or Chinese herbal medicine granules placebo — twice a day for 6 month
  Arms: Letrozole+ Chinese herbal medicine granules

SUMMARY:
This is a multicenter double-blind randomized controlled trial. A total of 420 anovulatory Chinese women with PCOS will be recruited, and the randomization will be stratified by each participating site. Participants will be randomized into one of the two treatment arms: letrozole and CHMG or letrozole and CHMG placebo. CHMG or its placebo will be taken twice a day for up to six months. Letrozole (2.5 mg daily) was given on days 3-7 of the menstrual cycle after a spontaneous period or withdrawal bleeding, and the dose will be increased to 5.0 mg daily during the last three months for non-pregnant women in both groups.The aim of the present study is to determine the efficacy of combined treatment with letrozole and CHMG on improving live birth rates in infertile Chinese women with PCOS. Our hypothesis is that the combination of letrozole and CHMG is more likely to increase the ovulation rate and decrease the miscarriage rate and result in a higher live birth rate in PCOS women than letrozole alone.

ELIGIBILITY:
Inclusion criteria

1. Chinese women with PCOS. PCOS must have been diagnosed based on the presence of two of the following three Rotterdam criteria : (1) oligomenorrhea, anovulation; (2) hyperandrogenism; and (3) the observation of polycystic ovaries by sonography. Oligomenorrhea is defined as an intermenstrual interval >35 days or <8 menstrual bleedings in the past year. Amenorrhea is defined as an intermenstrual interval >90 days.
2. History of at least one year of infertility.
3. Age between 20 and 40 years old.
4. Normal semen analysis based on World Health Organization criteria (2010). The husband did not need to sign the consent form because semen analysis is part of the clinical assessment at the sites. A sperm concentration ≥15 × 106/mL and total motility ≥40% in the semen analysis of the husband was required for the woman to be included.
5. Normal uterine cavity and at least one tube patent upon hysterosalpingography or HyCoSy.

Exclusion criteria

1. History of significant system diseases such as heart, lung, or kidney diseases.
2. History of other endocrine disorders.
3. Use of hormonal therapy, including metformin, in the past 3 months.
4. Previous sterilization procedures (vasectomy or tubal ligation) that have been reversed.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 420 (Estimated)
Dates: Start 2009-09; Primary Completion 2014-08 (Estimated); Study Completion 2014-08 (Estimated)

PRIMARY OUTCOMES:
Live birth rate | Up to 2 years

SECONDARY OUTCOMES:
Ovulation rate | Up to 1 year
Miscarriage rate | Up to 1 year
Change in hormonal profile | Up to 1 year
  Follicle-stimulating hormone, luteinizing hormone, total testosterone, sex hormone binding globulin, and dehydroepiandrosterone sulphate.
Change in metabolic profile | Up to 1 year
  glucose and insulin concentrations, cholesterol, triglycerides, high-density lipoprotein cholesterol and low-density lipoprotein cholesterol.
Change in physical measurements | Up to 1 year
  weight, vital signs, and hip and waist measurements.
Pregnancy complications | Up to 1 year
  gestational diabetes, pregnancy-induced hypertension, intrauterine growth retardation, ectopic pregnancy, congenital anomaly, preeclampsia, preterm labor, HELLP syndrome, preterm premature rupture of membranes, placental abruption, placenta accreta, placenta previa, postpartum hemorrhage, and others.
Birth defects | Up to 1 year
Safety parameters | Up to 1 year
  renal and liver function tests and complete blood count.
Side effect profile | Up to 1 year
  The major risks to the subject are side effects from letrozole and CHMG and the risks associated with pregnancy.

CONTACTS AND LOCATIONS:
Locations (18):
- China (18):
  - Affiliated Hospital of Anhui University of Chinese Medicine, Hefei, Anhui
  - Guangzhou Medical School First Affiliated Hospital, Guangzhou, Guangdong
  - Daqing Longnan hospital, Daqing, Heilongjiang
  - Daqing Oilfield General Hospital, Daqing, Heilongjiang
  - First Affliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - Dept Obs & Gyn, First Affiliated Hospital National Key Discipline and Trial Base Heilongjiang University of Chinese Medicine, Herbin, Heilongjiang
  - Mudanjiang maternal and children hospital, Mudanjiang, Heilongjiang
  - 2nd Affiliated Hospital of Henan University of Chinese Medicine, Zhengzhou, Henan
  - First Affiliated Hospital of Hunan University of Chinese, Changsha, Hunan
  - SuqianMaternal and Child Health Hospital, Suqian, Jiangsu
  - Maternal and Child Health Hospital of Xuzhou, Xuzhou, Jiangsu
  - First Hospital, Jiangxi college of Chinese Medicine, Nanchang, Jiangxi
  - Dalian Maternal and Child Health Hospital, Dalian, Liaoning
  - Shanxi Hospital of Chinese Medicine, Taiyuan, Shanxi
  - First Affiliated Hospital of Tianjin University of Chinese Medicine, Tianjin, Tianjin Municipality
  - Second Affiliated Hospital, Tianjin University of Chinese Medicine, Tianjin, Tianjin Municipality
  - Zhejiang province hospital of integrated traditional and western medicine, Hangzhou, Zhejiang
  - Second Affiliated Hospital of Heilongjiang University of Chinese Medicine, Harbin